CLINICAL TRIAL: NCT05846308
Title: The Effectiveness of Group Interpersonal Synchrony in Young Autistic Adults' Work Environment: A Mixed Methods RCT
Brief Title: The Effectiveness of Group Interpersonal Synchrony in Young Autistic Adults' Work Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Tal-Chen Rabinowitch, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2595
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Interpersonal Synchrony; Prosociality; work-related stress; Social closeness; Sense of belonging; Need to belong
MeSH Terms: conditions — Autism Spectrum Disorder; Occupational Stress

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized into one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous condition (Active Comparator): This arm (n=30) will include a synchronous intervention only.
  Interventions: Behavioral: Structured synchronous physical training
- Non-synchronous condition (Active Comparator): This arm (n=30) will include a non-synchronous intervention only.
  Interventions: Behavioral: Structured non-synchronous physical training

INTERVENTIONS:
Behavioral: Structured synchronous physical training — The instructors and the participants will form a circle facing each other while doing the physical exercises. To facilitate interpersonal synchrony, the participants will be instructed to do the same physical exercises (spatial synchrony) together at the same pace (rhythmic synchrony). Each session will consist of four parts:
  1. Warm-up (10 minutes)
  2. Social Game (10 minutes)
  3. Main training (30 minutes): Each session will contain two sets, each consisting of seven fixed exercises with a resting period of 10-15 seconds between each. Each exercise will be performed at one of three different paces: Slow - one movement cycle per 2 seconds, Medium - one movement cycle per 1 second and Fast - two movement cycles per 1 second.
  4. Cool-down (10 minutes)
  Arms: Synchronous condition
Behavioral: Structured non-synchronous physical training — The participants will do the same physical exercises as the participants in the synchronous group but in the form of circuit training with seven stations. The circuit training will require the participants to do a different physical exercise at a different pace at each station. A detailed description of the exercises will be provided for each station. The instructors will demonstrate all the exercises before the beginning of training. The participants will be instructed to do the exercise for a set period of time, the same duration used in the synchronous group. The circuit training stations will be in the form of a circle but will be set up so that the participants do not to face each other when doing the exercises to prevent spontaneous synchronization. Each session will consist of four parts, the same as in the synchronous intervention.
  Arms: Non-synchronous condition

SUMMARY:
Background: Few autistic adults are able to integrate successfully into the world of work given their difficulties adapting to the social and stressful aspects of work environments. Interpersonal synchrony, when two or more individuals share body movements or sensations, is a powerful force that consolidates human groups while promoting the ability to self-regulate and cooperate with others. The abilities to self-regulate and cooperate are crucial for maintaining a calm and productive work environment.

Objectives: This randomized controlled trial (RCT) aims to assess the effects of group interpersonal synchrony on prosociality and work-related stress of young autistic adults in their work environment.

Methods: This mixed-methods RCT will investigate two movement-based group synchronous and non-synchronous intervention conditions. The sample will be composed of young adults enrolled in an innovative Israeli program designed to integrate cognitively-abled 18- to 25-year-old autistic adults into the Israeli army work force. The movement-based intervention sessions will take place in groups of 10-14 participants, once a week for 10 weeks. Questionnaires, behavioral collaborative tasks and semi-structured interviews will be conducted. Quantitative data will be collected for each participant at three points of time: before and after the intervention period, and four months after the end of the intervention. Qualitative data will be collected after the intervention period in interviews with 15% of the participants.

DETAILED DESCRIPTION:
Background: Few autistic adults are able to integrate successfully into the world of work given their difficulties adapting to the social and stressful aspects of work environments. Interpersonal synchrony, when two or more individuals share body movements or sensations, is a powerful force that consolidates human groups while promoting the ability to self-regulate and cooperate with others. The abilities to self-regulate and cooperate are crucial for maintaining a calm and productive work environment.

Objectives: The objectives are to determine:

1. whether a synchronized group intervention will have an immediate and/or long-term positive effect on participants' prosociality and work-related stress.
2. whether this effect will be mediated by participants' reported social closeness and sense of belonging.
3. whether this effect will be influenced by participants' need to belong as reported before the intervention.
4. how participants perceive the intervention as affecting their prosociality and work-related stress.
5. in what ways the participants' perception of the intervention as affecting their prosociality and work-related stress will contribute to a better understanding of the intervention effect.

Methods: A mixed methods approach will be applied, where quantitative and qualitative data are collected and analyzed in parallel.

Participants: The sample will be composed of young adults (n=60) enrolled in an innovative Israeli program designed to integrate cognitively-abled 18- to 25-year-old autistic adults into the Israeli army workforce.

Sample Size: An a-priori power analysis indicated that a total sample size of 42 participants would be needed to detect medium effects defined as f=0.2, with 80% power and alpha at .05, using a repeated measure, within-between interaction ANOVA. This sample size might not be sufficient for detecting the mediated effect needed to respond to the second study objective with 80% power and alpha of .05. Therefore, we will recruit at least N = 60 participants (30 in each intervention group) to plan for possible dropouts.

Study Design and Procedures: This is a two-arm, randomized controlled trial (RCT) in which participants will be randomly assigned to one of two groups: synchronous and non-synchronous movement-based interventions. The movement-based intervention sessions will take place in groups of 10-14 participants, once a week for 10 weeks. A structured physical training protocol will be used for each condition. Each protocol is composed of 10 physical training sessions, each lasting 60 minutes. The protocols differ in terms of using synchronous activity vs. non-synchronous activity. They do not differ in terms of physical exercise type or duration to control for the effect of exercise type and duration on the dependent variables. Questionnaires, behavioral collaborative tasks and semi-structured interviews will be conducted. Quantitative data will be collected for each participant at three points of time: before and after the intervention period, and four months after the end of the intervention. Qualitative data will be collected after the intervention period in interviews with 15% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Trainees must have an official diagnosis of an autism spectrum disorder as assessed by a child psychiatrist or clinical psychologist according to the DSM-V.

Exclusion Criteria:

* Trainees with severe sensory impairments such as blindness or deafness and/or severe physical disability.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Work-related stress during baseline | Up to 1 month before start of intervention
  Work-related stress will be measured using the Hebrew adaptation of the Irritation Scale. This scale comprises eight items, three of which assess cognitive irritation and five of which assess emotional irritation. Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7).
Work-related stress during post-intervention | Up to 1 month after end of intervention
  Work-related stress will be measured using the Hebrew adaptation of the Irritation Scale. This scale comprises eight items, three of which assess cognitive irritation and five of which assess emotional irritation. Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7).
Work-related stress during follow-up | Between 3-4 month after end of intervention
  Work-related stress will be measured using the Hebrew adaptation of the Irritation Scale. This scale comprises eight items, three of which assess cognitive irritation and five of which assess emotional irritation. Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7).
Cognitive cooperation during baseline | Up to 1 month before start of intervention
  Cognitive cooperation will be measured using the Public Good Game task: Participants will be told they will be given 30 NIS and that they can donate some or all of it to a group investment. The money in the group investment will then be doubled and divided equally among all members of the group. Cooperation on this task will be operationalized by the amount of money each participant decides to donate to the group investment.
Cognitive cooperation during post-intervention | Up to 1 month after end of intervention
  Cognitive cooperation will be measured using the Public Good Game task: Participants will be told they will be given 30 NIS and that they can donate some or all of it to a group investment. The money in the group investment will then be doubled and divided equally among all members of the group. Cooperation on this task will be operationalized by the amount of money each participant decides to donate to the group investment.
Cognitive cooperation during follow-up | Between 3-4 month after end of intervention
  Cognitive cooperation will be measured using the Public Good Game task: Participants will be told they will be given 30 NIS and that they can donate some or all of it to a group investment. The money in the group investment will then be doubled and divided equally among all members of the group. Cooperation on this task will be operationalized by the amount of money each participant decides to donate to the group investment.
Behavioral cooperation during baseline | Up to 1 month before start of intervention
  Behavioral cooperation will be measured using the Collection task: Participants will have to work together to pick up 100 small washers (a flat plastic coin with a diameter of 4 cm). Cooperation on this task will be operationalized by participants' effort represented by their step rate (SR). SR will be measured using a wearable fitness tracker (Fitbit Inspire 2) that will be attached to the participants' wrists using a special band.
Behavioral cooperation during post-intervention | Up to 1 month after end of intervention
  Behavioral cooperation will be measured using the Collection task: Participants will have to work together to pick up 100 small washers (a flat plastic coin with a diameter of 4 cm). Cooperation on this task will be operationalized by participants' effort represented by their step rate (SR). SR will be measured using a wearable fitness tracker (Fitbit Inspire 2) that will be attached to the participants' wrists using a special band.
Behavioral cooperation during follow-up | Between 3-4 month after end of intervention
  Behavioral cooperation will be measured using the Collection task: Participants will have to work together to pick up 100 small washers (a flat plastic coin with a diameter of 4 cm). Cooperation on this task will be operationalized by participants' effort represented by their step rate (SR). SR will be measured using a wearable fitness tracker (Fitbit Inspire 2) that will be attached to the participants' wrists using a special band.

SECONDARY OUTCOMES:
Social Closeness during baseline | Up to 1 month before start of intervention
  Social Closeness will be measured using the Inclusion of Other in Self Scale. This scale is made up of seven Venn diagram-like pictures where one circle represents the participant and the other circle represents the entire intervention group.
Social Closeness during post-intervention | Up to 1 month after end of intervention
  Social Closeness will be measured using the Inclusion of Other in Self Scale. This scale is made up of seven Venn diagram-like pictures where one circle represents the participant and the other circle represents the entire intervention group.
Social Closeness during follow-up | Between 3-4 month after end of intervention
  Social Closeness will be measured using the Inclusion of Other in Self Scale. This scale is made up of seven Venn diagram-like pictures where one circle represents the participant and the other circle represents the entire intervention group.
Friendship Closeness during baseline | Up to 1 month before start of intervention
  Friendship Closeness will be measured using the Hebrew adaptation of the Friendship Closeness Inventory (FCI). The FCI is composed of 49 items that measure closeness in same-sex friendships and is divided into three distinguishable yet related subscales: Emotional Closeness (EC), Behavioral Closeness (BC), and Cognitive Closeness (CC). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the first item will be adjusted to include a reference to participants in the intervention group alone.
Friendship Closeness during post-intervention | Up to 1 month after end of intervention
  Friendship Closeness will be measured using the Hebrew adaptation of the Friendship Closeness Inventory (FCI). The FCI is composed of 49 items that measure closeness in same-sex friendships and is divided into three distinguishable yet related subscales: Emotional Closeness (EC), Behavioral Closeness (BC), and Cognitive Closeness (CC). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the first item will be adjusted to include a reference to participants in the intervention group alone.
Friendship Closeness during follow-up | Between 3-4 month after end of intervention
  Friendship Closeness will be measured using the Hebrew adaptation of the Friendship Closeness Inventory (FCI). The FCI is composed of 49 items that measure closeness in same-sex friendships and is divided into three distinguishable yet related subscales: Emotional Closeness (EC), Behavioral Closeness (BC), and Cognitive Closeness (CC). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the first item will be adjusted to include a reference to participants in the intervention group alone.
Sense of Belonging during baseline | Up to 1 month before start of intervention
  Sense of belonging will be measured using the Hebrew adaptation of the General Sense of Belonging Scale. This scale is composed of 12 items that measure sense of belonging (achieved belongingness). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the scale will be adjusted so that the words "other people" or "others" will be replaced by the words "participants in the physical training group".
Sense of Belonging during post-intervention | Up to 1 month after end of intervention
  Sense of belonging will be measured using the Hebrew adaptation of the General Sense of Belonging Scale. This scale is composed of 12 items that measure sense of belonging (achieved belongingness). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the scale will be adjusted so that the words "other people" or "others" will be replaced by the words "participants in the physical training group".
Sense of Belonging during follow-up | Between 3-4 month after end of intervention
  Sense of belonging will be measured using the Hebrew adaptation of the General Sense of Belonging Scale. This scale is composed of 12 items that measure sense of belonging (achieved belongingness). Items are rated on a 7-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7). For the purposes of this study, the scale will be adjusted so that the words "other people" or "others" will be replaced by the words "participants in the physical training group".
Need to Belong during baseline | Up to 1 month before start of intervention
  Need to Belong will be measured using the Hebrew adaptation of the Need to Belong Scale. This scale is composed of ten items rated on a 5-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (5).
Need to Belong during post-intervention | Up to 1 month after end of intervention
  Need to Belong will be measured using the Hebrew adaptation of the Need to Belong Scale. This scale is composed of ten items rated on a 5-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (5).
Need to Belong during follow-up | Between 3-4 month after end of intervention
  Need to Belong will be measured using the Hebrew adaptation of the Need to Belong Scale. This scale is composed of ten items rated on a 5-point Likert scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (5).

CONTACTS AND LOCATIONS:
Overall Officials: Tal-Chen Rabinowitch, PhD, Principal Investigator — University of Haifa, Israel
Locations (1):
- Roim Rachok Program, Or Yehuda, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dvir T, Elefant C, Rabinowitch TC. Group Interpersonal Synchrony Increases Prosocial Behavior in Young Autistic Adults: A Randomized Controlled Trial. J Autism Dev Disord. 2025 Jul 5. doi: 10.1007/s10803-025-06949-y. Online ahead of print. PMID 40615734
- [Derived] Dvir T, Rabinowitch TC, Elefant C. The effectiveness of group interpersonal synchrony in young autistic adults' work environment: A mixed methods RCT study protocol. PLoS One. 2024 Jul 31;19(7):e0307956. doi: 10.1371/journal.pone.0307956. eCollection 2024. PMID 39083478